CLINICAL TRIAL: NCT02163694
Title: A Phase 3 Randomized, Placebo-Controlled Trial of Carboplatin and Paclitaxel With or Without the PARP Inhibitor Veliparib (ABT-888) in HER2-Negative Metastatic or Locally Advanced Unresectable BRCA-Associated Breast Cancer
Brief Title: A Phase 3 Randomized, Placebo-controlled Trial of Carboplatin and Paclitaxel With or Without Veliparib (ABT-888) in HER2-negative Metastatic or Locally Advanced Unresectable BRCA-associated Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12-914; 2014-000345-70 (EudraCT Number)
Record Dates: First submitted 2014-05-19; First posted 2014-06-16 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Breast Cancer
Keywords: PARP Inhibitor; Veliparib; BRCA1; BRCA2; HER2-negative; Locally recurrent; Breast Cancer; Metastatic Breast Cancer; ABT-888; Genetic breast cancer; Paclitaxel; BRCA Mutation; PARP; Carboplatin; BROCADE3
MeSH Terms: conditions — Breast Neoplasms | interventions — veliparib; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veliparib Placebo with Carboplatin and Paclitaxel (Active Comparator): Placebo capsules for veliparib (120 mg) administered by mouth twice daily (BID) on Days -2 through 5 of a 21-day cycle. Carboplatin administered intravenously over approximately 15 to 30 minutes at AUC 6 mg/ml/min immediately following paclitaxel infusion on Day 1 of every cycle. Paclitaxel administered intravenously over approximately 1 hour at a dose of 80 mg/m² on Days 1, 8, and 15 of every cycle.
  Interventions: Drug: Veliparib Placebo; Drug: Carboplatin; Drug: Paclitaxel
- Veliparib with Carboplatin and Paclitaxel (Experimental): Veliparib capsules (120 mg) administered by mouth twice daily (BID) on Days -2 through 5 of a 21-day cycle. Carboplatin administered intravenously over approximately 15 to 30 minutes at AUC 6 mg/ml/min immediately following paclitaxel infusion on Day 1 of every cycle. Paclitaxel administered intravenously over approximately 1 hour at a dose of 80 mg/m² on Days 1, 8, and 15 of every cycle.
  Interventions: Drug: Veliparib; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Veliparib Placebo — Supplied as 40 mg, 50 mg, or 100 mg capsules for oral administration twice daily (BID) on Days -2 through 5 of a 21-day cycle.
  Arms: Veliparib Placebo with Carboplatin and Paclitaxel
Drug: Veliparib — Supplied as 40 mg, 50 mg, or 100 mg capsules for oral administration twice daily (BID) on Days -2 through 5 of a 21-day cycle.
  Other Names: ABT-888
  Arms: Veliparib with Carboplatin and Paclitaxel
Drug: Carboplatin — Administered intravenously over approximately 15 to 30 minutes at an area under the curve (AUC) of 6 mg/mL/min immediately following paclitaxel infusion on Day 1 of every cycle. The duration of carboplatin infusion may be lengthened according to institutional guidelines.
Drug: Paclitaxel — Administered by intravenous infusion over approximately 1 hour at a dose of 80 mg/m² of body-surface area (BSA) on Days 1, 8, and 15 of each 21-day cycle. Paclitaxel is to be infused prior to carboplatin on Day 1. Dosing of veliparib/placebo is to be completed before the carboplatin or paclitaxel infusions.

SUMMARY:
The primary objective of the study is to assess the progression-free survival (PFS) of veliparib in combination with carboplatin and paclitaxel (C/P) compared to placebo plus C/P in participants with a Breast Cancer Gene 1 or 2 (BRCA1; BRCA2) mutation in Human Epidermal Growth Factor Receptor 2 (HER2)-negative metastatic or locally advanced unresectable breast cancer. The secondary objectives of the study are to assess overall survival (OS), clinical benefit rate (CBR) through the end of Week 24, objective response rate (ORR) and PFS on subsequent therapy (PFS2) in participants treated with veliparib in combination with C/P versus placebo in combination with C/P.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, multinational, multicenter study to evaluate the efficacy and tolerability of veliparib in combination with C/P compared to placebo in combination with C/P in participants with a BRCA1 or BRCA2 mutation, as documented by the Sponsor core laboratory, with HER2-negative metastatic or locally advanced unresectable breast cancer who received no more than 2 prior lines of cytotoxic therapy for metastatic disease. For the purposes of eligibility, HER2-negative status was based on the most recent tumor biopsy. Participants were randomized in a 2:1 ratio, with a total of approximately 500 participants planned to be randomized. Veliparib 120 mg/placebo twice a day (BID) was dosed Days -2 through 5 with carboplatin target area under the concentration-time curve (AUC) 6 administered on Day 1 and paclitaxel 80 mg/m2 administered weekly on Days 1, 8, and 15 of each 21-day cycle.

Safety and efficacy data through the prespecified primary analysis cutoff date of 05 April 2019 are included in the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed breast cancer that is either locally advanced or metastatic. Locally advanced breast cancer must not be amenable to surgical resection or radiation with curative intent.
2. Suspected deleterious or deleterious Breast Cancer Gene 1 (BRCA1) and/or Breast Cancer Gene 2 (BRCA2) germline mutation.
3. Breast cancer must be Human Epidermal Growth Factor Receptor 2 (HER2)-negative.
4. Measurable or non-measurable (but radiologically evaluable) disease per Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1 on computed tomography (CT) scan (within 28 days of randomization) with at least one lesion outside previously irradiated areas.
5. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 2.
6. Adequate hematologic, renal, and hepatic function (within 28 days of randomization).

Exclusion Criteria:

1. More than two prior lines of cytotoxic chemotherapy (e.g., gemcitabine, doxorubicin, capecitabine) for metastatic disease.

   * Regimens received in the adjuvant/neoadjuvant setting or for locally advanced breast cancer within the past 6 months will also be considered toward the maximum of 2 prior lines of therapy. Adjuvant/neoadjuvant chemotherapy for one cancer event will count as one prior line of therapy, if received within the past 6 months.
   * Previous treatments with hormonal therapy (tamoxifen, aromatase inhibitors) and signal transduction agents (e.g., erlotinib, gefitinib, everolimus, bevacizumab) are allowed and are not counted towards the prior line of therapy.
2. Progressed or recurred within 12 months of completing platinum therapy or received > 1 prior line of platinum therapy for breast cancer in any setting (adjuvant, neoadjuvant, or metastatic).
3. Prior therapy with Poly(ADP-ribose)-Polymerase (PARP) inhibitors.
4. Prior taxane therapy administered for the treatment of metastatic breast cancer with the below exceptions.

   * Prior taxane therapy for metastatic breast cancer is allowed if the patient received ≤ 1 full cycle (i.e., therapy discontinued within 4 weeks for subjects receiving weekly paclitaxel or Abraxane; therapy discontinued within 3 weeks for subjects receiving paclitaxel or docetaxel every 3 weeks) in the absence of progression or if taxane therapy for metastatic disease was > 12 months prior to Cycle 1 Day-2 (C1D-2).
   * Use of taxanes as adjuvant therapy or to treat locally advanced disease is permitted, if given more than 6 months prior to C1D-2
5. Known history of allergic reaction to cremophor-paclitaxel, carboplatin, Azo-Colourant Tartrazine (also known as FD&C Yellow 5 or E102), Azo-Colourant Orange Yellow-S (also known as FD&C Yellow 6 or E110) or known contraindications to any study supplied drug.
6. Active CNS metastases or leptomeningeal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (219):
- United States (56):
  - Banner MD Anderson Cancer Ctr /ID# 125011, Gilbert, Arizona
  - University of Arkansas for Medical Sciences /ID# 124992, Little Rock, Arkansas
  - City of Hope /ID# 127117, Duarte, California
  - California Cancer Associates for Research & Excellence (cCARE) /ID# 136078, Fresno, California
  - Moores Cancer Center at UC San Diego /ID# 124991, La Jolla, California
  - Hematology and Oncology Assoc /ID# 130058, Newport Beach, California
  - Cancer Research Collaboration /ID# 128860, Santa Ana, California
  - Icri /Id# 128520, Whittier, California
  - Univ of Colorado Cancer Center /ID# 124983, Aurora, Colorado
  - Saint Joseph Hospital /ID# 131768, Denver, Colorado
  - Norwalk Hospital /ID# 133509, Norwalk, Connecticut
  - Lynn Cancer Institute, Boca /ID# 125013, Boca Raton, Florida
  - Holy Cross Hospital /ID# 125012, Fort Lauderdale, Florida
  - Sacred Heart Hospital /ID# 128279, Pensacola, Florida
  - Moffitt Cancer Center /ID# 124990, Tampa, Florida
  - Florida Cancer Specialists - East /ID# 125007, West Palm Beach, Florida
  - Emory Midtown Infectious Disease Clinic /ID# 133192, Atlanta, Georgia
  - The Cancer Ctr at DeKalb Med C /ID# 125024, Decatur, Georgia
  - University of Illinois - Chicago /ID# 127576, Chicago, Illinois
  - NorthShore University HealthSystem /ID# 124996, Evanston, Illinois
  - Midwestern Regional CTC /ID# 124986, Zion, Illinois
  - McFarland Clinic, PC /ID# 129904, Ames, Iowa
  - Johns Hopkins University /ID# 125015, Baltimore, Maryland
  - Baystate Medical Center /ID# 139461, Springfield, Massachusetts
  - UMass Chan Medical School /ID# 129067, Worcester, Massachusetts
  - Henry Ford Health System /ID# 134497, Detroit, Michigan
  - Spectrum Health Medical Group /ID# 133568, Grand Rapids, Michigan
  - Spectrum Health Medical Group /ID# 148471, Grand Rapids, Michigan
  - William Beaumont Hospital /ID# 125019, Royal Oak, Michigan
  - Univ of Mississippi Med Ctr,US /ID# 131352, Jackson, Mississippi
  - St. Lukes Cancer Institute /ID# 125023, Kansas City, Missouri
  - Washington University-School of Medicine /ID# 127575, St Louis, Missouri
  - Nebraska Hematology Oncology /ID# 132711, Lincoln, Nebraska
  - Rutgers Cancer Institute of New Jersey /ID# 125017, New Brunswick, New Jersey
  - University of New Mexico /ID# 125349, Albuquerque, New Mexico
  - Beth Israel Medical Center /ID# 125001, New York, New York
  - Mount Sinai St. Luke's /ID# 125003, New York, New York
  - Mission Cancer Center /ID# 134248, Asheville, North Carolina
  - Duke Cancer Center /ID# 124999, Durham, North Carolina
  - The Ohio State University /ID# 125022, Columbus, Ohio
  - University of Toledo /ID# 134849, Toledo, Ohio
  - Oregon Health and Science University /ID# 134229, Portland, Oregon
  - Lehigh Valley Health Network /ID# 130059, Allentown, Pennsylvania
  - Lehigh Valley Hosp/Muhlenberg /ID# 130277, Bethlehem, Pennsylvania
  - Penn State University and Milton S. Hershey Medical Center /ID# 124997, Hershey, Pennsylvania
  - Allegheny General Hospital /ID# 135094, Pittsburgh, Pennsylvania
  - University of Pittsburgh MC /ID# 125005, Pittsburgh, Pennsylvania
  - Texas Health Physicians Group /ID# 137740, Arlington, Texas
  - University of Texas Southwestern Medical Center /ID# 124989, Dallas, Texas
  - University of Texas MD Anderson Cancer Center /ID# 125353, Houston, Texas
  - University of Vermont Medical Center /ID# 125350, Burlington, Vermont
  - Swedish Cancer Institute - Issaquah /ID# 131534, Issaquah, Washington
  - Swedish Cancer Institute - Edmonds /ID# 131549, Seattle, Washington
  - Swedish Medical Center /ID# 125021, Seattle, Washington
  - Swedish Cancer Insititute - Ballard /ID# 131548, Seattle, Washington
  - Northwest Medical Specialties - Tacoma /ID# 125344, Tacoma, Washington
- Argentina (4):
  - COIBA Centro de Oncologia e Investigacion de Buenos Aires /ID# 124839, Berazategui, Buenos Aires
  - Clinica Pergamino /ID# 127158, Pergamino, Buenos Aires
  - Instituto de Oncoloia de Rosario /ID# 127157, Rosario, Santa Fe Province
  - Centro Oncologico Riojano Integral /ID# 127938, La Rioja
- Australia (8):
  - St George Hospital /ID# 129416, Kogarah, New South Wales
  - Duplicate_The Prince of Wales Hospital /ID# 124845, Randwick, New South Wales
  - Southern Medical Day Care Centre /ID# 124844, Wollongong, New South Wales
  - Townsville University Hospital /ID# 126731, Douglas, Queensland
  - Duplicate_Flinders Centre for Innovation /ID# 127535, Bedford Park, South Australia
  - Royal Hobart Hospital /ID# 124849, Hobart, Tasmania
  - The Royal Melbourne Hospital /ID# 124846, Parkville, Victoria
  - Hollywood Private Hospital /ID# 124843, Nedlands, Western Australia
- Austria (4):
  - Medizinische Universitaet Graz /ID# 126450, Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 126185, Linz, Upper Austria
  - Medizinische Universitaet Wien /ID# 126184, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitätsklinikum der PMU (LKH) /ID# 126449, Salzburg
- Belarus (4):
  - Bobruysk Interdistrict Onco. /ID# 137729, Babruysk
  - State Institution Republican Scientific Practical Center of Oncology and Medical /ID# 125223, Minsk
  - Duplicate_Mogilev Reg Clin Oncology Dis /ID# 137728, Mogilev
  - Vitebsk Regional Clinical Oncology Dispensary /ID# 125219, Vitebsk
- Belgium (7):
  - Universitair Ziekenhuis Antwerpen /ID# 124977, Edegem, Antwerpen
  - UCL Saint-Luc /ID# 124976, Woluwe-Saint-Lambert, Brussels Capital
  - Grand Hôpital de Charleroi /ID# 124981, Charleroi, Hainaut
  - Universitair Ziekenhuis Leuven /ID# 124980, Leuven, Vlaams-Brabant
  - Duplicate_AZ St-Jan Brugge-Oostende AV /ID# 124975, Bruges, West-Vlaanderen
  - ZNA Middelheim /ID# 124978, Antwerp
  - CHU UCL Namur - Sainte Elisabeth /ID# 124979, Namur
- Canada (4):
  - Duplicate_Sunnybrook Health Sciences Ctr /ID# 124882, Toronto, Ontario
  - CHUM - Notre-Dame Hospital /ID# 124879, Montreal, Quebec
  - Duplicate_Jewish General Hospital /ID# 124880, Montreal, Quebec
  - Duplicate_CHUQ-Hospital St. Sacrement /ID# 124881, Québec, Quebec
- Chile (4):
  - Hospital Clinico Vina del Mar /ID# 130100, Viña del Mar, Región de Valparaíso
  - Hospital Clinico Vina del Mar /ID# 148502, Viña del Mar, Región de Valparaíso
  - Instituto Nacional del Cancer /ID# 129343, Santiago
  - ICOS - Inst Clinic Oncology /ID# 125236, Temuco
- Colombia (5):
  - Hospital Pablo Tobon Uribe /ID# 126657, Medellín, Antioquia
  - Administradora del Country_S.A-Clinica Del Country /ID# 125255, Bogota, Cundinamarca
  - Hospital Univ San Ignacio /ID# 126655, Bogota, Cundinamarca
  - Instituto Medico de Alta Tecnologia Oncomédica S.A /ID# 129211, Montería, Departamento de Córdoba
  - Centro Medico Imbanaco de Cali /ID# 126656, Cali
- Czechia (5):
  - Fakultni Nemocnice Brno /ID# 128176, Brno
  - Masarykuv onkologicky ustav /ID# 124886, Brno
  - Duplicate_FN Hradec Kralove /ID# 127080, Hradec Králové
  - Fakultni nemocnice Olomouc /ID# 124885, Olomouc
  - Vseobecna fakultni nemocnice v Praze /ID# 124887, Prague
- Denmark (2):
  - Rigshospitalet /ID# 124891, Copenhagen Ø, Capital Region
  - Sygehus Lillebælt, Vejle /ID# 124892, Vejle, Region Syddanmark
- East Tallinn Central Hospital /ID# 126475, Kesklinn, Harju, Estonia
- Finland (4):
  - Docrates Cancer Center /ID# 124896, Helsinki
  - Duplicate_Helsinki Univ Central Hospital /ID# 124897, Helsinki
  - Duplicate_Tampere University Hospital /ID# 124898, Tampere
  - Vaasa Central Hospital /ID# 132548, Vaasa
- France (4):
  - Institut Paoli-Calmettes /ID# 124903, Marseille, Bouches-du-Rhone
  - Institut de Cancérologie de l'Ouest René Gauducheau /ID# 137726, Saint-Herblain, Loire-Atlantique
  - Institut Curie - site CLCC René Huguenin /ID# 124904, Saint-Cloud
  - Institut Curie /ID# 124902, Paris, Île-de-France Region
- Germany (7):
  - Universitaetsklinik Heidelberg /ID# 126664, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinimum Tuebingen /ID# 129968, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 135230, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Koeln /ID# 126905, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 127180, Dresden
  - Klinikum rechts der Isar - Technische Universitaet Muenchen /ID# 125256, Munich
  - Sana Klinikum Offenbach /ID# 126733, Offenbach
- Hungary (4):
  - Semmelweis Egyetem /ID# 132485, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 125259, Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz /ID# 124911, Szolnok
  - Duplicate_Zala Megyei Korhaz /ID# 131341, Zalaegerszeg
- Israel (8):
  - The Chaim Sheba Medical Center /ID# 124918, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 130276, Tel Aviv, Tel Aviv
  - Duplicate_Soroka University Medical Center /ID# 124917, Beersheba
  - Assaf Harofeh Medical Center /ID# 124915, Be’er Ya‘aqov
  - Rambam Health Care Campus /ID# 124916, Haifa
  - Shaare Zedek Medical Center /ID# 130275, Jerusalem
  - Gastroenterology Institute, Division of Medicine /ID# 124919, Jerusalem
  - Kaplan Medical Center /ID# 124914, Rehovot
- Italy (5):
  - Ospedale San Raffaele IRCCS /ID# 125261, Milan, Lombardy
  - IEO -Istituto Europeo di Oncologia /ID# 125260, Milan, Milano
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 125262, Negrar, Verona
  - Centro di Riferimento Oncologico /ID# 126738, Aviano
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli /ID# 125263, Reggio Calabria
- Latvia (2):
  - Pauls Stradins Clinical University Hospital /ID# 125264, Riga
  - Riga East Clinical University Hospital /ID# 125265, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 125266, Kaunas
  - National Cancer Institute /ID# 125267, Vilnius
- Mexico (3):
  - Centro de Estudios Clínicos Especializados /ID# 128680, Mérida, Yucatán
  - Centro Oncologico de Chihuahua /ID# 128679, Chihuahua City
  - Instituto Nacional de Cancerología INCAN /ID# 128676, Mexico City
- Netherlands (3):
  - Erasmus Medisch Centrum /ID# 124935, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen /ID# 129069, Groningen
  - Maastricht Universitair Medisch Centrum /ID# 129068, Maastricht
- Haukeland University Hospital /ID# 150177, Bergen, Hordaland, Norway
- Poland (5):
  - Centrum Onkologii Lukaszczyka /ID# 124938, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalistyczny /ID# 127258, Wroclaw, Lower Silesian Voivodeship
  - MRUK-MED I Spolka z ograniczona odpowiedzialnoscia /ID# 124939, Rzeszów, Podkarpackie Voivodeship
  - Wojewodzki Szpital Zespolony /ID# 126998, Elblag, Warmian-Masurian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopern /ID# 126999, Lodz, Łódź Voivodeship
- Portugal (6):
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE /ID# 126510, Vila Nova de Gaia, Porto District
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital Faro /ID# 125298, Faro
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 125299, Lisbon
  - Unidade Local de Saúde de Matosinhos, EPE /ID# 126511, Matosinhos Municipality
  - IPO Porto FG, EPE /ID# 125297, Porto
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 126508, Porto
- Puerto Rico (2):
  - Ad-Vance Medical Research, LLC /ID# 126043, Ponce
  - San Juan Municipal Hospital /ID# 124695, San Juan
- Romania (4):
  - S.C. Centrul de Oncologie Sf. Nectarie S.R.L. /ID# 124948, Craiova, Dolj
  - Duplicate_lnstitutul Oncologic Prof Dr Alexandru Trestioreanu /ID# 124943, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj -Napoca /ID# 124945, Cluj-Napoca
  - Oncomed SRL /ID# 127598, Timișoara
- Russia (9):
  - Sverdlovsk Regional Oncology Dispensary /ID# 130950, Yekaterinburg, Sverdlovsk Oblast
  - Regional Oncology Dispensary /ID# 125936, Kursk, Tatarstan, Respublika
  - Duplicate_archangel Clinical Oncology /ID# 126031, Arkhangelsk
  - Altay Regional Oncological Dispesary /ID# 127160, Barnaul
  - Belgorod Oncology Dispensary /ID# 129315, Belgorod
  - LLC BioEq Ltd. /ID# 134529, Saint Petersburg
  - Duplicate_Saratov State Medical University n.s. Chernyshevskiy /ID# 139395, Saratov
  - Siberian State Medical University /ID# 127161, Tomsk
  - Volgograd Regional Clinical Oncology Dispensary /ID# 124952, Volzhsky
- Singapore (2):
  - National University Hospital /ID# 125315, Singapore
  - Johns Hopkins Singapore IMC /ID# 125316, Singapore
- South Africa (9):
  - GVI Oncology /ID# 125321, Port Elizabeth, Eastern Cape
  - University of Free State, Universitas Annex (National Hospital Grounds) /ID# 128499, Bloemfontein, Free State
  - Wits Clinical Research Site /ID# 125317, Johannesburg, Gauteng
  - Medical Oncology Ctr Rosebank /ID# 125322, Johannesburg, Gauteng
  - Sandton Oncology Medical Group PTY Ltd /ID# 125323, Johannesburg, Gauteng
  - Mary Potter Oncology Centre /ID# 133269, Pretoria, Gauteng
  - The Oncology Centre /ID# 126104, Durban, KwaZulu-Natal
  - Netcare Oncology Intervent Ctr /ID# 125320, Cape Town, Western Cape
  - Cancercare Outeniqua Oncology Centre /ID# 125319, George, Western Cape
- South Korea (6):
  - National Cancer Center /ID# 125602, Goyang, Gyeonggido
  - Yonsei University Health System Severance Hospital /ID# 125599, Seoul, Seoul Teugbyeolsi
  - Korea University Anam Hospital /ID# 128968, Seoul
  - Seoul National University Hospital /ID# 125600, Seoul
  - Asan Medical Center /ID# 125601, Seoul
  - Samsung Medical Center /ID# 125598, Seoul
- Spain (5):
  - Hospital Santa Creu i Sant Pau /ID# 124963, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 124962, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 124960, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 124961, Málaga
  - Hospital Clinico Universitario de Valencia /ID# 124959, Valencia
- Sweden (6):
  - Skane University hospital /ID# 124966, Malmo, Skåne County
  - Norrlands University hospital /ID# 124967, Umeå, Västerbotten County
  - Sahlgrenska University Hospital /ID# 124965, Gothenburg, Västra Götaland County
  - Linkoping University Hospital /ID# 126795, Linköping
  - Duplicate_Karolinska Univ Sjukhuset /ID# 124964, Solna
  - Uppsala University Hospital /ID# 126512, Uppsala
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 125575, Kaohsiung City
  - National Taiwan University Hospital /ID# 125324, Taipei
- Turkey (Türkiye) (5):
  - Hacettepe University Faculty of Medicine /ID# 125336, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi /ID# 125337, Ankara
  - Duplicate_Akdeniz University Medical Fac /ID# 125339, Antalya
  - Bezmi Alem Univ Med Fac Hosp /ID# 127901, Istanbul
  - Istanbul University Istanbul Medical Faculty /ID# 145144, Istanbul
- Ukraine (7):
  - Municipal Non-Profit Enterprise City Clinical Hospital No.4 of Dnipro City Counc /ID# 124968, Dnipro
  - Donetsk Regional Antitumor Ctr /ID# 124970, Donetsk
  - Communal non-profit enterprise Regional Center of Oncology /ID# 124972, Kharkiv
  - ME Kryviy Rih Oncology Dispensary /ID# 129806, Kryvyi Rih
  - Lviv Oncological Regional Therapeutical and Diagnostic Centre /ID# 124974, Lviv
  - Poltava Regional Clinical Oncology Centre of Poltava Regional Council /ID# 124969, Poltava
  - Zaporizhzhia Med. Academy MOH /ID# 129800, Zaporizhia
- United Kingdom (4):
  - University Hospitals Bristol /ID# 128343, Bristol, Bristol, City of
  - Hull University Teaching Hospitals NHS Trust /ID# 133030, Hull, East Riding Of Yorkshire
  - Nottingham University Hospitals NHS Trust /ID# 125340, Nottingham, Nottinghamshire
  - University Hospitals Birmingham NHS Foundation Trust /ID# 125342, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Stodtmann S, Eckert D, Joshi R, Nuthalapati S, Ratajczak CK, Menon R, Mensing S, Xiong H. Exposure-Response Model With Time-Varying Predictors to Estimate the Effects of Veliparib in Combination With Carboplatin/Paclitaxel and as Monotherapy: Veliparib Phase 3 Study in BRCA-Mutated Advanced Breast Cancer (BROCADE3) Trial. J Clin Pharmacol. 2022 Oct;62(10):1236-1246. doi: 10.1002/jcph.2061. Epub 2022 May 5. PMID 35403245
- [Derived] Ayoub JP, Wildiers H, Friedlander M, Arun BK, Han HS, Puhalla S, Shparyk Y, Jakobsen EH, Wu M, Bach BA, Feng D, Ratajczak CK, Maag D, Dieras V. Safety and efficacy of veliparib plus carboplatin/paclitaxel in patients with HER2-negative metastatic or locally advanced breast cancer: subgroup analyses by germline BRCA1/2 mutations and hormone receptor status from the phase-3 BROCADE3 trial. Ther Adv Med Oncol. 2021 Dec 9;13:17588359211059601. doi: 10.1177/17588359211059601. eCollection 2021. PMID 34917174
- [Derived] Arun BK, Han HS, Kaufman B, Wildiers H, Friedlander M, Ayoub JP, Puhalla SL, Bell-McGuinn KM, Bach BA, Kundu MG, Ratajczak CK, Maag D, Dieras V. Efficacy and safety of first-line veliparib and carboplatin-paclitaxel in patients with HER2- advanced germline BRCA+ breast cancer: Subgroup analysis of a randomised clinical trial. Eur J Cancer. 2021 Sep;154:35-45. doi: 10.1016/j.ejca.2021.05.037. Epub 2021 Jul 6. PMID 34243076
- [Derived] Puhalla SL, Dieras V, Arun BK, Kaufman B, Wildiers H, Han HS, Ayoub JP, Stearns V, Yuan Y, Helsten T, Riley-Gillis B, Murphy E, Kundu MG, Wu M, Maag D, Ratajczak CK, Ramathal CY, Friedlander M. Relevance of Platinum-free Interval and BRCA Reversion Mutations for Veliparib Monotherapy after Progression on Carboplatin/Paclitaxel for gBRCA Advanced Breast Cancer (BROCADE3 Crossover). Clin Cancer Res. 2021 Sep 15;27(18):4983-4993. doi: 10.1158/1078-0432.CCR-21-0748. Epub 2021 Jun 15. PMID 34131001
- [Derived] Dieras V, Han HS, Kaufman B, Wildiers H, Friedlander M, Ayoub JP, Puhalla SL, Bondarenko I, Campone M, Jakobsen EH, Jalving M, Oprean C, Palacova M, Park YH, Shparyk Y, Yanez E, Khandelwal N, Kundu MG, Dudley M, Ratajczak CK, Maag D, Arun BK. Veliparib with carboplatin and paclitaxel in BRCA-mutated advanced breast cancer (BROCADE3): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Oct;21(10):1269-1282. doi: 10.1016/S1470-2045(20)30447-2. Epub 2020 Aug 27. PMID 32861273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 513 subjects enrolled in the study (N=174 to the placebo + C/P arm, and N=339 to the veliparib + C/P arm). Two subjects form each arm (N= 4) were determined not to have a suspected deleterious or deleterious mutation in BRCA1/2 and were excluded from the ITT population [ITT Population (N=509); Placebo + C/P arm (N=172), and Veliparib + C/P arm (N=337)]. Of the 4 subjects, 3 subjects received treatment and later discontinued due to disease progression.
Pre-assignment Details: Subjects randomized to placebo were eligible to crossover to unblinded veliparib monotherapy. After Protocol Amendment 5, investigators and subjects were unblinded to treatment assignment, subjects randomized to placebo discontinued from the study, subjects discontinuing therapy prior to progression no longer remained on study, and no new subjects initiated crossover unblinded veliparib monotherapy treatment.
Groups:
- Placebo + C/P: Placebo capsules for veliparib (120 mg) administered by mouth twice daily (BID) on Days -2 through 5 of a 21-day cycle. Carboplatin administered intravenously over approximately 15 to 30 minutes at AUC 6 mg/ml/min immediately following paclitaxel infusion on Day 1 of every cycle. Paclitaxel administered intravenously over approximately 1 hour at a dose of 80 mg/m² on Days 1, 8, and 15 of every cycle.
- Veliparib + C/P: Veliparib capsules (120 mg) administered by mouth twice daily (BID) on Days -2 through 5 of a 21-day cycle. Carboplatin administered intravenously over approximately 15 to 30 minutes at AUC 6 mg/ml/min immediately following paclitaxel infusion on Day 1 of every cycle. Paclitaxel administered intravenously over approximately 1 hour at a dose of 80 mg/m² on Days 1, 8, and 15 of every cycle.
Period: Overall Study
Arm/Group | Placebo + C/P | Veliparib + C/P
Started | 174 | 339
ITT Population | 172 | 337
Completed | 0 | 0
Not Completed | 174 | 339
Not completed — Adverse event- related to progression | 4 | 10
Not completed — Adverse event- not related to progression | 7 | 22
Not completed — Withdrew consent | 13 | 28
Not completed — Lost to Follow-up | 2 | 2
Not completed — Sponsor discontinued study | 3 | 29
Not completed — Progressive disease per protocol | 125 | 224
Not completed — Other, not specified | 17 | 22
Not completed — Randomized but Not Treated | 1 | 0
Not completed — Determined not to have a suspected deleterious or deleterious mutation in BRCA1/2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + C/P | Veliparib + C/P | Total
Number analyzed (Participants) | 172 | 337 | 509
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (10.81) | 46.8 (10.73) | 46.8 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 333 | 502
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 153 | 294 | 447
  Black or African American | 6 | 14 | 20
  Asian | 12 | 24 | 36
  American Indian or Alaska Native | 0 | 3 | 3
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Multiple | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Time to PFS is defined as the number of days from the date the participant was randomized to the date the participant experiences radiographic disease progression (as determined by the investigators), or to the date of death (all causes of mortality) if disease progression is not reached. All events of disease progression occurring on or before the Primary Analysis Cutoff date of 05 April 2019 were to be included, regardless of whether the event occurred while the participant was still taking study drug or had previously discontinued study drug. PFS was estimated for each treatment group using Kaplan-Meier methodology.
Time Frame: From randomization until the primary analysis data cut-off date of 05 April 2019; the median duration of follow-up was 35.5 months
Population: ITT population for whom data was collected and available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + C/P | Veliparib + C/P
Number analyzed (Participants) | 172 | 337
months | 12.6 [10.6 to 14.4] | 14.6 [12.5 to 17.7]
Statistical Analysis 1: Comparison: Placebo + C/P vs Veliparib + C/P; PFS was compared between the treatment groups using the log-rank test, stratified by prior platinum therapy (Yes versus No) and receptor status (estrogen receptor [ER] and/or progesterone receptor [PgR] positive versus ER/PgR negative); Test type: Superiority; p = 0.003, Log-rank test
Statistical Analysis 2: Comparison: Placebo + C/P vs Veliparib + C/P; A Cox proportional hazards model, stratified by prior platinum therapy (Yes versus No) and receptor status (estrogen receptor (ER) and/or progesterone receptor (PgR) positive versus ER/PgR negative) was used to estimate the hazard ratio and 95% confidence interval comparing the two treatment arms; Test type: Superiority; p = 0.003, Stratified Cox proportional hazards; Stratified Cox proportional hazards = 0.728, 95% CI 2-sided [0.590 to 0.900]

2. Secondary Outcome: Overall Survival (OS)
Description: Time to death (overall survival) is defined as the number of days from the date the participant was randomized to the date of the participant's death. All events of death which occur up to the analysis cutoff date are to be included, regardless of whether the event occurred while the participant was still taking study drug or after the participant discontinued study drug. If a participant has not died, the data for the participant is to be censored at the date last known to be alive or at the analysis cutoff date if that is earlier.
  The final analysis of OS will occur when the pre-specified number of events has occurred in the ITT population.
Time Frame: Up to 84.5 and 81.8 months for Placebo and Veliparib, respectively.
Population: ITT population for whom data was collected and available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + C/P | Veliparib + C/P
Number analyzed (Participants) | 172 | 337
months | 28.2 [24.7 to 32.8] | 32.4 [27.4 to 38.1]
Statistical Analysis 1: Comparison: Placebo + C/P vs Veliparib + C/P; Test type: Superiority; p = 0.410, Log Rank
Statistical Analysis 2: Comparison: Placebo + C/P vs Veliparib + C/P; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.410, Stratified Cox proportional hazards; Stratified Cox proportional hazards = 0.914, 95% CI 2-sided [0.737 to 1.333]

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The clinical benefit rate (CBR) is defined as the progression-free rate at 24 weeks (168 days), estimated using Kaplan Meier methodology. All events of disease progression in the primary progression free survival analysis database were to be included, regardless of whether the event occurred while the participant was still taking, or had previously discontinued, study drug. If the participant had not yet progressed then their data was to be censored at the date of the last evaluable disease progression assessment. Participants without post-baseline assessments were to be censored at the date of randomization.
Time Frame: Through the end of Week 24
Population: ITT population for whom data was collected and available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + C/P | Veliparib + C/P
Number analyzed (Participants) | 172 | 337
percentage of participants | 93.2 [89.5 to 95.7] | 90.7 [87.9 to 92.9]
Statistical Analysis 1: Comparison: Placebo + C/P vs Veliparib + C/P; Test type: Superiority; p = 0.202, Cochran-Mantel-Haenszel — Nominal P value is from Cochran-Mantel-Haenszel test stratified by ER/PgR status and prior platinum therapy use

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The objective response rate (ORR) is calculated as the percentage of participants who have a confirmed partial response (PR) or complete response (CR) based on assessment by the investigators per Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1. All participants who had at least one measurable lesion at baseline were to be included in the ORR calculation.
  The final analysis of ORR will occur when the pre-specified number of Overall Survival events have occurred in the ITT population, per the fixed sequence testing procedure.
Time Frame: Approximately 8 years from randomization
Population: ITT population for whom data was collected and available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + C/P | Veliparib + C/P
Number analyzed (Participants) | 172 | 337
percentage of participants | 74.1 [66.1 to 81.1] | 75.8 [70.4 to 80.6]
Statistical Analysis 1: Comparison: Placebo + C/P vs Veliparib + C/P; Test type: Superiority; p = 0.715, Cochran-Mantel-Haenszel — Nominal P value is from Cochran-Mantel-Haenszel test stratified by ER/PgR status and prior platinum therapy use

5. Secondary Outcome: Progression-Free Survival on Subsequent Therapy (PFS2)
Description: PFS2 is defined as the number of days from the date of randomization to the time of disease progression on subsequent therapy or death from any cause. The distribution of PFS2 was to be estimated for each treatment group using Kaplan-Meier methodology.
  The final analysis of PFS2 will occur when the pre-specified number of Overall Survival events have occurred in the ITT population, per the fixed sequence testing procedure.
Time Frame: Approximately 8 years from randomization
Population: ITT population for whom data was collected and available for analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + C/P | Veliparib + C/P
Number analyzed (Participants) | 172 | 337
months | 17.4 [16.0 to 20.7] | 21.5 [19.9 to 25.3]
Statistical Analysis 1: Comparison: Placebo + C/P vs Veliparib + C/P; Test type: Superiority; p = 0.004, Log Rank
Statistical Analysis 2: Comparison: Placebo + C/P vs Veliparib + C/P; Test type: Superiority; p = 0.004, Stratified Cox proportional hazards; Stratified by prior platinum therapy (yes vs no) and receptor status (ER and/or PgR positive vs ER/PgR negative); Stratified Cox proportional hazards = 0.737, 95% CI 2-sided [0.597 to 0.908]

ADVERSE EVENTS:
Time Frame: All-cause mortality were reported from enrollment to the end of study, median time on follow up was 84.5 and 81.8 months for Placebo + C/P and Veliparib + C/P, respectively. Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 30 days after the last dose of study drug; mean duration on study drug was 115.0 and 117.5 days for Placebo + C/P and Veliparib + C/P, respectively.
Groups:
- Placebo + C/P: Placebo capsules for veliparib (120 mg) administered by mouth twice daily (BID) on Days -2 through 5 of a 21- day cycle. Carboplatin administered intravenously over approximately 15 to 30 minutes at AUC 6 mg/ml/min immediately following paclitaxel infusion on Day 1 of every cycle. Paclitaxel administered intravenously over approximately 1 hour at a dose of 80 mg/m² on Days 1, 8, and 15 of every cycle.
Arm/Group | Placebo + C/P | Veliparib + C/P
All-Cause Mortality (participants affected / at risk) | 129/174 | 244/339
Serious Adverse Events (participants affected / at risk) | 68/174 | 135/339
Other Adverse Events (participants affected / at risk) | 169/174 | 332/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + C/P (N=174) | Veliparib + C/P (N=339)
ANAEMIA (Blood and lymphatic system disorders) | 5 (9) | 16 (21)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 11 (11)
HAEMORRHAGIC DISORDER (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 8 (11)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 (7) | 14 (21)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (4)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1)
RETINAL ARTERY OCCLUSION (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS MICROSCOPIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 2 (3)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 2 (2)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 6 (9)
NONINFECTIVE SIALOADENITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 6 (8)
CHEST PAIN (General disorders) | 1 (1) | 3 (3)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 2 (4)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0)
HYPERTHERMIA (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 1 (1)
PAIN (General disorders) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 4 (5) | 9 (12)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 2 (2)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 2 (2)
CONTRAST MEDIA ALLERGY (Immune system disorders) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 3 (3) | 1 (1)
HAEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS (Immune system disorders) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
ABSCESS JAW (Infections and infestations) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 2 (2)
BREAST CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS MORAXELLA (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 4 (5)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (2)
ERYSIPELAS (Infections and infestations) | 2 (2) | 2 (3)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
INFECTED DERMAL CYST (Infections and infestations) | 0 (0) | 1 (1)
INFECTED LYMPHOCELE (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 2 (4) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 3 (3)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
MENINGITIS (Infections and infestations) | 1 (1) | 0 (0)
MYELITIS (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1)
NEUTROPENIC INFECTION (Infections and infestations) | 0 (0) | 2 (2)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
PAROTID ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 1 (2)
PNEUMONIA (Infections and infestations) | 2 (2) | 7 (8)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 4 (4) | 4 (4)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 3 (3)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (3)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 2 (2) | 5 (5)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
JOINT LOCK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (6)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 19 (26)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO BONE MARROW (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (7)
SECOND PRIMARY MALIGNANCY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
APHASIA (Nervous system disorders) | 0 (0) | 1 (1)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 2 (3)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CERVICAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 2 (2)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0)
INTRACRANIAL PRESSURE INCREASED (Nervous system disorders) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
MENINGEAL DISORDER (Nervous system disorders) | 0 (0) | 1 (2)
PARTIAL SEIZURES (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 1 (1) | 1 (1)
SEIZURE (Nervous system disorders) | 2 (2) | 4 (4)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
DEVICE BREAKAGE (Product Issues) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 1 (1)
MANIA (Psychiatric disorders) | 1 (1) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (2)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY ARTERY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 (3) | 1 (1)
ILIAC ARTERY OCCLUSION (Vascular disorders) | 0 (0) | 1 (1)
POOR VENOUS ACCESS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + C/P (N=174) | Veliparib + C/P (N=339)
ANAEMIA (Blood and lymphatic system disorders) | 117 (501) | 256 (1147)
LEUKOPENIA (Blood and lymphatic system disorders) | 65 (319) | 133 (700)
LYMPHOPENIA (Blood and lymphatic system disorders) | 14 (33) | 43 (139)
NEUTROPENIA (Blood and lymphatic system disorders) | 156 (1286) | 292 (2450)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 118 (581) | 257 (1659)
PALPITATIONS (Cardiac disorders) | 4 (4) | 20 (28)
TACHYCARDIA (Cardiac disorders) | 11 (16) | 14 (20)
TINNITUS (Ear and labyrinth disorders) | 8 (8) | 21 (43)
VERTIGO (Ear and labyrinth disorders) | 14 (20) | 24 (38)
DRY EYE (Eye disorders) | 10 (11) | 24 (26)
VISION BLURRED (Eye disorders) | 9 (10) | 10 (13)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 7 (10) | 18 (19)
ABDOMINAL PAIN (Gastrointestinal disorders) | 24 (30) | 52 (81)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 23 (33) | 56 (90)
CONSTIPATION (Gastrointestinal disorders) | 59 (87) | 117 (183)
DIARRHOEA (Gastrointestinal disorders) | 69 (141) | 151 (337)
DRY MOUTH (Gastrointestinal disorders) | 17 (17) | 34 (42)
DYSPEPSIA (Gastrointestinal disorders) | 20 (24) | 61 (88)
GASTRITIS (Gastrointestinal disorders) | 10 (10) | 4 (5)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 8 (8) | 18 (20)
NAUSEA (Gastrointestinal disorders) | 118 (328) | 240 (772)
STOMATITIS (Gastrointestinal disorders) | 24 (32) | 46 (74)
TOOTHACHE (Gastrointestinal disorders) | 11 (12) | 26 (30)
VOMITING (Gastrointestinal disorders) | 72 (160) | 118 (280)
ASTHENIA (General disorders) | 45 (141) | 85 (346)
CHEST PAIN (General disorders) | 14 (15) | 19 (29)
FATIGUE (General disorders) | 90 (218) | 168 (383)
INFLUENZA LIKE ILLNESS (General disorders) | 15 (26) | 27 (50)
MUCOSAL INFLAMMATION (General disorders) | 7 (7) | 30 (37)
OEDEMA PERIPHERAL (General disorders) | 20 (25) | 69 (96)
PAIN (General disorders) | 11 (11) | 20 (22)
PERIPHERAL SWELLING (General disorders) | 9 (10) | 18 (21)
PYREXIA (General disorders) | 35 (45) | 59 (83)
DRUG HYPERSENSITIVITY (Immune system disorders) | 32 (66) | 58 (91)
BRONCHITIS (Infections and infestations) | 5 (6) | 21 (27)
INFLUENZA (Infections and infestations) | 7 (7) | 19 (26)
NASOPHARYNGITIS (Infections and infestations) | 27 (42) | 60 (89)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (5) | 17 (26)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 10 (16) | 15 (33)
RHINITIS (Infections and infestations) | 4 (5) | 20 (24)
SINUSITIS (Infections and infestations) | 9 (12) | 29 (34)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 19 (27) | 52 (86)
URINARY TRACT INFECTION (Infections and infestations) | 17 (43) | 41 (77)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 25 (61) | 59 (151)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 23 (62) | 50 (115)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 9 (18) | 26 (48)
WEIGHT INCREASED (Investigations) | 5 (13) | 19 (40)
DECREASED APPETITE (Metabolism and nutrition disorders) | 56 (71) | 81 (106)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (4) | 17 (23)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 9 (19) | 22 (65)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 14 (21) | 29 (55)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 19 (47) | 44 (95)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 39 (108) | 83 (196)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 (5) | 18 (24)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 9 (28) | 26 (51)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 58 (98) | 77 (133)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 42 (62) | 66 (105)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 23 (39) | 41 (54)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 9 (13) | 20 (25)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 9 (9) | 25 (29)
MYALGIA (Musculoskeletal and connective tissue disorders) | 26 (39) | 60 (88)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 8 (11) | 17 (23)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 40 (53) | 71 (119)
DIZZINESS (Nervous system disorders) | 34 (53) | 68 (114)
DYSGEUSIA (Nervous system disorders) | 19 (27) | 48 (61)
HEADACHE (Nervous system disorders) | 67 (113) | 124 (217)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 15 (19) | 22 (27)
PARAESTHESIA (Nervous system disorders) | 16 (30) | 33 (40)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 89 (185) | 158 (347)
TASTE DISORDER (Nervous system disorders) | 13 (19) | 19 (39)
ANXIETY (Psychiatric disorders) | 13 (17) | 40 (48)
DEPRESSION (Psychiatric disorders) | 10 (12) | 30 (36)
INSOMNIA (Psychiatric disorders) | 33 (47) | 63 (84)
BREAST PAIN (Reproductive system and breast disorders) | 10 (13) | 19 (25)
COUGH (Respiratory, thoracic and mediastinal disorders) | 34 (48) | 77 (126)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 34 (43) | 71 (105)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 7 (18) | 24 (32)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 29 (37) | 62 (87)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 31 (44)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 18 (23)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 21 (29)
ALOPECIA (Skin and subcutaneous tissue disorders) | 87 (113) | 182 (254)
DRY SKIN (Skin and subcutaneous tissue disorders) | 6 (7) | 27 (29)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 9 (18) | 18 (20)
PRURITUS (Skin and subcutaneous tissue disorders) | 8 (12) | 32 (45)
RASH (Skin and subcutaneous tissue disorders) | 22 (28) | 43 (58)
HOT FLUSH (Vascular disorders) | 13 (16) | 41 (52)
HYPERTENSION (Vascular disorders) | 12 (14) | 25 (40)
LYMPHOEDEMA (Vascular disorders) | 11 (15) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT02163694/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT02163694/SAP_001.pdf